CLINICAL TRIAL: NCT05319418
Title: PILOT: Effectiveness of BP Remote Monitoring Software With Virtual Physician Management in Stage 2 Hypertension Patients With History of Stroke or TIA.
Brief Title: Effectiveness of BP Remote Monitoring With Virtual Physician Management in Hypertensive Patients.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: AIRx Health, Inc. (Other)
Collaborators: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 61821
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Hypertension; Stroke (CVA) or TIA
Keywords: remote patient monitoring; digital health monitoring; blood pressure monitoring
MeSH Terms: conditions — Hypertension; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hypertensive Patients Monitored Daily (Experimental): Physicians utilize DailyDoctor remote monitoring platform to virtually monitor daily BP of patients. Physicians use their independent medical judgement to recommend any clinical follow up or adjustment in medications/prescriptions for any patients whose daily reporting of BP triggers an alert based on physician-driven alert thresholds.
  Interventions: Behavioral: Daily Blood Pressure Monitoring

INTERVENTIONS:
Behavioral: Daily Blood Pressure Monitoring — Patients are provided standard off-the-shelf blood pressure monitors and take their BP vitals daily. Patients report their daily BP through phone or online. BP data is viewed online by physicians who use their independent medical judgement for any changes in medical management.

SUMMARY:
To assess the feasibility and adoptability of DailyDoctor's remote monitoring clinical decision support software tool in helping physicians virtually manage systolic blood pressures among patients with history of stroke or TIA to a target systolic blood pressure (<140 mmHg or a lower target range specified by referring physicians) using remote monitoring and independent clinical judgement.

DETAILED DESCRIPTION:
To assess the feasibility and adoptability of DailyDoctor's remote monitoring clinical decision support software tool in helping physicians virtually manage systolic blood pressures among patients with history of stroke or TIA to a target systolic blood pressure (<140 mmHg or a lower target range specified by referring physicians) using remote monitoring and independent clinical judgement.

To assess the feasibility and adoptability of DailyDoctor's digital platform in helping Stanford Stroke Center lower and maintain systolic blood pressures among patients with history of stroke or TIA to a target systolic blood pressure (<140 mmHg or a lower target range specified by referring physicians) using remote monitoring and a virtual medical team focused on BP management.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older. A history of ischemic or hemorrhagic stroke, or transient ischemic attack. The ability to report blood pressure values by phone (either a patient or designated caregiver may call to report values).

At least 2 BP measurements that are ≥140 mmHg systolic or ≥90 mmHg diastolic obtained on different days in the last 6 months in any setting (including at home, in clinic, or in the hospital setting).

The referring physician feels the patient would benefit from BP optimization. Consent to receive care from telehealth physicians available through the DailyDoctor monitoring platform.

English or Spanish speaking.

Exclusion Criteria:

Currently enrolled in another interventional research study Inability to comply with study protocol Have a planned surgical procedure during the study period Upper arm circumference > 20 inches Has diagnosis of end-stage renal disease (GFR < 15 mL/min), Serum creatinine > 2.0 mg/dL (176.8 μmol/L), or currently undergoing dialysis treatment (10) Women who are pregnant or who are planning to become pregnant during the study period.

Blood pressure reduction is not indicated (e.g. patients who have a high blood pressure target to augment cerebral perfusion).

Any other reason that, in the opinion of the investigator, makes the person a poor candidate for participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Percent patients within target BP | 24 Weeks
  The change in the percentage of patients who are within their target blood pressure range between baseline (based on the average of the first 5 BP readings recorded by the patient using the DailyDoctor platform) and at the completion of the 24 week interv

SECONDARY OUTCOMES:
Change in average systolic blood pressure | 24 Weeks
  The average systolic blood pressure of the first 5 BP readings recorded by a patient using the DailyDoctor platform will be compared to the average of the last 5 readings of systolic blood pressure reported by the patient using the DailyDoctor platform.
Proportion of patients within target BP range | Every 4-week period over 24 weeks.
  Proportions of patients who are within their target blood pressure range during every 4-week period over 24 weeks.
Time taken to achieve a clinically significant reduction in blood pressure | Varies, recorded over 24 weeks
  Time taken to achieve a clinically significant reduction in blood pressure (5mmHg for systolic blood pressure or 2.5 mmHg in diastolic blood pressure)
Participant compliance | Recorded over 24 weeks
  Participant compliance, defined as the percentage of days that a patient transmits a vital sign reading on a monthly or weekly basis.
Rate of blood pressure decline | Recorded over 24 weeks
  Rate of blood pressure decline
Change in number of antihypertensive drugs | 24 Weeks
  Change in number of antihypertensive drugs prescribed between baseline and the final assessment
Change in number of classes of antihypertensive drugs | 24 Weeks
  Change in number of classes of antihypertensive drugs prescribed between baseline and the final assessment with 5 predefined classes: diuretics, angiotensin-converting enzyme inhibitors and angiotensin receptor blockers, calcium channel blockers, β-blockers, and others (α-blockers, hydralazine, minoxidil, clonidine, reserpine, guanethidine, and methyldopa).
Number and types of AEs & SAEs | Recorded over 24 weeks
  Number and types of AEs & SAEs
Proportions of patients of various BP categories | Recorded over 24 weeks
  Based on weekly and 4-weekly blood pressure averages, the proportions of patients who are classified as:
  Normal (<120 mmHg systolic/ <80 mmHg diastolic) Elevated (120-129 mmHg systolic/ <80 mmHg diastolic). Stage 1 hypertensive: systolic pressure ranging from 130 to 139 mm Hg or a diastolic pressure ranging from 80 to 89 mm Hg.
  Stage 2 hypertensive: systolic pressure ≥140 mm Hg or a diastolic pressure ≥90 mm Hg.

CONTACTS AND LOCATIONS:
Overall Officials: Maarten Lansberg, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford Stroke Center, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kitagawa K, Yamamoto Y, Arima H, Maeda T, Sunami N, Kanzawa T, Eguchi K, Kamiyama K, Minematsu K, Ueda S, Rakugi H, Ohya Y, Kohro T, Yonemoto K, Okada Y, Higaki J, Tanahashi N, Kimura G, Umemura S, Matsumoto M, Shimamoto K, Ito S, Saruta T, Shimada K; Recurrent Stroke Prevention Clinical Outcome (RESPECT) Study Group. Effect of Standard vs Intensive Blood Pressure Control on the Risk of Recurrent Stroke: A Randomized Clinical Trial and Meta-analysis. JAMA Neurol. 2019 Nov 1;76(11):1309-1318. doi: 10.1001/jamaneurol.2019.2167. PMID 31355878
- [Background] Spruill TM, Williams O, Teresi JA, Lehrer S, Pezzin L, Waddy SP, Lazar RM, Williams SK, Jean-Louis G, Ravenell J, Penesetti S, Favate A, Flores J, Henry KA, Kleiman A, Levine SR, Sinert R, Smith TY, Stern M, Valsamis H, Ogedegbe G. Comparative effectiveness of home blood pressure telemonitoring (HBPTM) plus nurse case management versus HBPTM alone among Black and Hispanic stroke survivors: study protocol for a randomized controlled trial. Trials. 2015 Mar 15;16:97. doi: 10.1186/s13063-015-0605-5. PMID 25873044
- [Background] SPRINT Research Group; Wright JT Jr, Williamson JD, Whelton PK, Snyder JK, Sink KM, Rocco MV, Reboussin DM, Rahman M, Oparil S, Lewis CE, Kimmel PL, Johnson KC, Goff DC Jr, Fine LJ, Cutler JA, Cushman WC, Cheung AK, Ambrosius WT. A Randomized Trial of Intensive versus Standard Blood-Pressure Control. N Engl J Med. 2015 Nov 26;373(22):2103-16. doi: 10.1056/NEJMoa1511939. Epub 2015 Nov 9. PMID 26551272
- [Background] Ho TW, Huang CT, Chiu HC, Ruan SY, Tsai YJ, Yu CJ, Lai F; HINT Study Group. Effectiveness of Telemonitoring in Patients with Chronic Obstructive Pulmonary Disease in Taiwan-A Randomized Controlled Trial. Sci Rep. 2016 Mar 31;6:23797. doi: 10.1038/srep23797. PMID 27029815
- [Background] Achelrod D, Schreyogg J, Stargardt T. Health-economic evaluation of home telemonitoring for COPD in Germany: evidence from a large population-based cohort. Eur J Health Econ. 2017 Sep;18(7):869-882. doi: 10.1007/s10198-016-0834-x. Epub 2016 Oct 3. PMID 27699567
- [Background] Weissman GE, Kerlin MP, Yuan Y, Kohn R, Anesi GL, Groeneveld PW, Werner RM, Halpern SD. Potentially Preventable Intensive Care Unit Admissions in the United States, 2006-2015. Ann Am Thorac Soc. 2020 Jan;17(1):81-88. doi: 10.1513/AnnalsATS.201905-366OC. PMID 31581801
- [Background] Logan AG, McIsaac WJ, Tisler A, Irvine MJ, Saunders A, Dunai A, Rizo CA, Feig DS, Hamill M, Trudel M, Cafazzo JA. Mobile phone-based remote patient monitoring system for management of hypertension in diabetic patients. Am J Hypertens. 2007 Sep;20(9):942-8. doi: 10.1016/j.amjhyper.2007.03.020. PMID 17765133
- [Background] Stevens LA, Greene T, Levey AS. Surrogate end points for clinical trials of kidney disease progression. Clin J Am Soc Nephrol. 2006 Jul;1(4):874-84. doi: 10.2215/CJN.00600206. Epub 2006 Jun 14. No abstract available. PMID 17699300
- See also: Citation 14 — https://www.mgma.com/MGMA/media/files/fellowship%20papers/2018%20Fellows%20Papers/Neurology-Workforce-Shortage-KB-FACMPE-FINAL-9-20-2018.pdf?ext=.pdf